CLINICAL TRIAL: NCT04564677
Title: A Prospective Study Evaluating the Clinical Outcome of a Modified d'Hoore Technique for Laparoscopic Ventral Mesh Rectopexy
Brief Title: A Study Evaluating the Clinical Outcome of a Modified d'Hoore Technique for Laparoscopic Ventral Mesh Rectopexy
Acronym: POP-01
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Duomed (Industry)
Responsible Party: Sponsor
Other Study IDs: DM-ZOL-02
Record Dates: First submitted 2020-09-03; First posted 2020-09-25 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Rectocele; Enterocele; Rectal Prolapse
MeSH Terms: conditions — Rectocele; Hernia; Rectal Prolapse

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients eligible for laparoscopic ventral mesh rectopexy: Female patients with primary rectal prolapse, rectocele and/or enterocele eligible for laparoscopic ventral mesh rectopexy (LVMR)
  Interventions: Device: Ifabond (Péters surgical)

INTERVENTIONS:
Device: Ifabond (Péters surgical) — Ifabond (Péters surgical) is a CE-marked synthetic surgical glue for internal and external use. The glue is non-toxic, biocompatible and biodegradable. It is commercially available and can be used for mesh fixation, as tissue adhesive, for sealing of sutured tissue and for hemostasis.

SUMMARY:
The purpose of this observational study is to evaluate the clinical outcome of a modified d'Hoore technique for laparoscopic ventral mesh rectopexy in patients with primary rectal prolapse, rectocele and/or enterocele.The goal of the study will be achieved by reporting the peri- and postoperative complications ((serious) adverse events), recurrences and re-interventions. Pre-operative to postoperative changes in pain, functional outcome and quality of life will be evaluated as well.

ELIGIBILITY:
Inclusion Criteria:

* Female patients.
* Patient ≥ 18 years of age at study entry.
* Patient and investigator signed and dated the informed consent form prior to the index-procedure.
* Patient with primary rectal prolapse (grades I to V according to the Oxford scale), rectocele and/or enterocele.

Exclusion Criteria:

* Patient is unable / unwilling to provide informed consent.
* Patient with recurrent rectal prolapse, rectocele and/or enterocele.
* Patient is unable to comply with the study protocol or proposed follow-up visits.
* Patient has a contra-indication for laparoscopic ventral mesh rectopexy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients with primary rectal prolapse, rectocele and/or enterocele eligible for laparoscopic ventral mesh rectopexy.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-02-08 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Procedural efficacy - Number of participants with (serious) adverse events | During procedure
  Number of participants with (serious) adverse events ≥ grade II Clavien-Dindo
Procedural efficacy - Conversion rate to laparotomy during the index procedure | During procedure
  Number of conversions to laparotomy during the index procedure
Procedural efficacy - Number of participants with (serious) adverse events | At discharge (assessed up to 1 week)
  Number of participants with (serious) adverse events ≥ grade II Clavien-Dindo
Procedural efficacy - Number of re-interventions | At discharge (assessed up to 1 week)
  Number of re-interventions
Procedural efficacy - Number of participants with (serious) adverse events | Follow-up 1: 6 - 10 weeks after the procedure
  Number of participants with (serious) adverse events ≥ grade II Clavien-Dindo
Procedural efficacy - Number of re-interventions | Follow-up 1: 6 - 10 weeks after the procedure
  Number of re-interventions
Procedural efficacy - Number of post-operative recurrences | Follow-up 1: 6 - 10 weeks after the procedure
  Number of post-operative recurrences
Procedural efficacy - Number of participants with (serious) adverse events | Follow-up 2: 12 months after the procedure
  Number of participants with (serious) adverse events ≥ grade II Clavien-Dindo
Procedural efficacy - Number of re-interventions | Follow-up 2: 12 months after the procedure
  Number of re-interventions
Procedural efficacy - Number of post-operative recurrences | Follow-up 2: 12 months after the procedure
  Number of post-operative recurrences
Procedural efficacy - Number of participants with (serious) adverse events | Follow-up 3: 24 months after the procedure
  Number of participants with (serious) adverse events ≥ grade II Clavien-Dindo
Procedural efficacy - Number of re-interventions | Follow-up 3: 24 months after procedure
  Number of re-interventions
Procedural efficacy - Number of post-operative recurrences | Follow-up 3: 24 months after the procedure
  Number of post-operative recurrences
Procedural efficacy - Number of participants with (serious) adverse events | Follow-up 4: 36 months after the procedure
  Number of participants with (serious) adverse events ≥ grade II Clavien-Dindo
Procedural efficacy - Number of re-interventions | Follow-up 4: 36 months after the procedure
  Number of re-interventions
Procedural efficacy - Number of post-operative recurrences | Follow-up 4: 36 months after the procedure
  Number of post-operative recurrences

SECONDARY OUTCOMES:
Pre-operative abdominal pain by means of the Visual Analogue Scale (VAS) | At baseline
  Assessment of pre-operative abdominal pain by means of the VAS, which contains a 0 to 100 grading scale with 0 equaling no pain and 100 equaling the worst conceivable pain.
Pre-operative vaginal pain by means of the Visual Analogue Scale (VAS) | At baseline
  Assessment of pre-operative vaginal pain by means of the VAS, which contains a 0 to 100 grading scale with 0 equaling no pain and 100 equaling the worst conceivable pain.
Functional score - Obstructive Defecation Syndrome (ODS) score | At baseline
  The ODS score is obtained by means of a structured 8-item questionnaire on multiple bowel symptoms. The cumulative score for all answers ranges from 0 to 31, with higher scores being indicative of more severe symptoms.
Functional score - Cleveland Clinical Incontinence Score (CCIS) | At baseline
  The CCIS is a 5-item questionnaire used to score the level of fecal incontinence. The cumulative score ranges from 0 to 20, with higher scores being indicative of more severe symptoms.
Quality of life - Birmingham Bowel and Urinary Symptoms Questionnaire (BBUSQ) | At baseline
  The BBUSQ is a 22-item questionnaire to record data on 4 domains: constipation, evacuation, incontinence and urinary symptoms. Higher scores are indicative of more severe symptoms.
Post-operative abdominal pain by means of the Visual Analogue Scale (VAS) | Follow-up 1: 6 - 10 weeks after the procedure
  Assessment of post-operative abdominal pain by means of the VAS, which contains a 0 to 100 grading scale with 0 equaling no pain and 100 equaling the worst conceivable pain.
Post-operative abdominal pain by means of the Visual Analogue Scale (VAS) | Follow-up 2: 12 months after the procedure
  Assessment of post-operative abdominal pain by means of the VAS, which contains a 0 to 100 grading scale with 0 equaling no pain and 100 equaling the worst conceivable pain.
Post-operative abdominal pain by means of the Visual Analogue Scale (VAS) | Follow-up 3: 24 months after the procedure
  Assessment of post-operative abdominal pain by means of the VAS, which contains a 0 to 100 grading scale with 0 equaling no pain and 100 equaling the worst conceivable pain.
Post-operative abdominal pain by means of the Visual Analogue Scale (VAS) | Follow-up 4: 36 months after the procedure
  Assessment of post-operative abdominal pain by means of the VAS, which contains a 0 to 100 grading scale with 0 equaling no pain and 100 equaling the worst conceivable pain.
Post-operative vaginal pain by means of the Visual Analogue Scale (VAS) | Follow-up 1: 6 - 10 weeks after the procedure
  Assessment of post-operative vaginal pain by means of the VAS, which contains a 0 to 100 grading scale with 0 equaling no pain and 100 equaling the worst conceivable pain.
Post-operative vaginal pain by means of the Visual Analogue Scale (VAS) | Follow-up 2: 12 months after the procedure
  Assessment of post-operative vaginal pain by means of the VAS, which contains a 0 to 100 grading scale with 0 equaling no pain and 100 equaling the worst conceivable pain.
Post-operative vaginal pain by means of the Visual Analogue Scale (VAS) | Follow-up 3: 24 months after the procedure
  Assessment of post-operative vaginal pain by means of the VAS, which contains a 0 to 100 grading scale with 0 equaling no pain and 100 equaling the worst conceivable pain.
Post-operative vaginal pain by means of the Visual Analogue Scale (VAS) | Follow-up 4: 36 months after the procedure
  Assessment of post-operative vaginal pain by means of the VAS, which contains a 0 to 100 grading scale with 0 equaling no pain and 100 equaling the worst conceivable pain.
Functional score - Obstructive Defecation Syndrome (ODS) score | Follow-up 1: 6 - 10 weeks after the procedure
  The ODS score is obtained by means of a structured 8-item questionnaire on multiple bowel symptoms. The cumulative score for all answers ranges from 0 to 31, with higher scores being indicative of more severe symptoms.
Functional score - Obstructive Defecation Syndrome (ODS) score | Follow-up 2: 12 months after the procedure
  The ODS score is obtained by means of a structured 8-item questionnaire on multiple bowel symptoms. The cumulative score for all answers ranges from 0 to 31, with higher scores being indicative of more severe symptoms.
Functional score - Obstructive Defecation Syndrome (ODS) score | Follow-up 3: 24 months after the procedure
  The ODS score is obtained by means of a structured 8-item questionnaire on multiple bowel symptoms. The cumulative score for all answers ranges from 0 to 31, with higher scores being indicative of more severe symptoms.
Functional score - Obstructive Defecation Syndrome (ODS) score | Follow-up 4: 36 months after the procedure
  The ODS score is obtained by means of a structured 8-item questionnaire on multiple bowel symptoms. The cumulative score for all answers ranges from 0 to 31, with higher scores being indicative of more severe symptoms.
Functional score - Cleveland Clinical Incontinence Score (CCIS) | Follow-up 1: 6 - 10 weeks after the procedure
  The CCIS is a 5-item questionnaire used to score the level of fecal incontinence. The cumulative score ranges from 0 to 20, with higher scores being indicative of more severe symptoms.
Functional score - Cleveland Clinical Incontinence Score (CCIS) | Follow-up 2: 12 months after the procedure
  The CCIS is a 5-item questionnaire used to score the level of fecal incontinence. The cumulative score ranges from 0 to 20, with higher scores being indicative of more severe symptoms.
Functional score - Cleveland Clinical Incontinence Score (CCIS) | Follow-up 3: 24 months after the procedure
  The CCIS is a 5-item questionnaire used to score the level of fecal incontinence. The cumulative score ranges from 0 to 20, with higher scores being indicative of more severe symptoms.
Functional score - Cleveland Clinical Incontinence Score (CCIS) | Follow-up 4: 36 months after the procedure
  The CCIS is a 5-item questionnaire used to score the level of fecal incontinence. The cumulative score ranges from 0 to 20, with higher scores being indicative of more severe symptoms.
Quality of life - Birmingham Bowel and Urinary Symptoms Questionnaire (BBUSQ) | Follow-up 1: 6 - 10 weeks after the procedure
  The BBUSQ is a 22-item questionnaire to record data on 4 domains: constipation, evacuation, incontinence and urinary symptoms. Higher scores are indicative of more severe symptoms.
Quality of life - Birmingham Bowel and Urinary Symptoms Questionnaire (BBUSQ) | Follow-up 2: 12 months after the procedure
  The BBUSQ is a 22-item questionnaire to record data on 4 domains: constipation, evacuation, incontinence and urinart symptoms. Higher scores are indicative of more severe symptoms.
Quality of life - Birmingham Bowel and Urinary Symptoms Questionnaire (BBUSQ) | Follow-up 3: 24 months after the procedure
  The BBUSQ is a 22-item questionnaire to record data on 4 domains: constipation, evacuation, incontinence and urinary symptoms. Higher scores are indicative of more severe symptoms.
Quality of life - Birmingham Bowel and Urinary Symptoms Questionnaire (BBUSQ) | Follow-up 4: 36 months after the procedure
  The BBUSQ is a 22-item questionnaire to record data on 4 domains: constipation, evacuation, incontinence and urinary symptoms. Higher scores are indicative of more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Dams, MD, Principal Investigator — Ziekenhuis Oost-Limburg (ZOL)
Locations (1):
- Ziekenhuis Oost-Limburg (ZOL), Genk, Belgium

IPD SHARING:
Plan to Share IPD: No